CLINICAL TRIAL: NCT00752323
Title: Fluorescence-Guided Detection of Malignant Gliomas: A Dose Ranging Study Using 5-Aminolevulinic Acid (ALA) Induced Protoporphyrin (PpIX) in a Multicenter Phase II Clinical Trial
Brief Title: Imaging Procedure Using ALA in Finding Residual Tumor in Grade IV Malignant Astrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Sloan, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew Sloan, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CASE1305
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neurosurgeons and investigators responsible for determining pathologic characteristics, for quantifying fluorescence images, for extracting chemical PpIX, for co-localizing fluorescence images with MR images will be blinded to the ALA dose and administration time. In case of emergency, such as toxicity or allergic reaction attributable to the drug, the research pharmacist on call will break the blind and inform the physician responsible for clinical management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm I: Newly diagnosed GBM 10mg/kg (Experimental): Arm I: Newly diagnosed GBM patients receive oral aminolevulinic acid(10mg/kg)at 6 hours before the midpoint of surgery.
  Interventions: Drug: aminolevulinic acid; Procedure: Surgical Resection
- Arm II: Newly diagnosed GBM 20mg/kg (Experimental): Arm II: Newly diagnosed GBM patients receive oral aminolevulinic acid (20mg/kg)at 6 hours before the midpoint of surgery.
  Interventions: Drug: aminolevulinic acid; Procedure: Surgical Resection
- Arm III: Recurrent GBM 10mg/kg (Experimental): Arm III: Recurrent GBM patients receive oral aminolevulinic acid (10mg/kg)at 6 hours before the midpoint of surgery.
  Interventions: Drug: aminolevulinic acid; Procedure: Surgical Resection
- Arm IV: Recurrent GBM 20mg/kg (Experimental): Arm IV: Recurrent GBM patients receive oral aminolevulinic acid (20mg/kg)at 6 hours before the midpoint of surgery.
  Interventions: Drug: aminolevulinic acid; Procedure: Surgical Resection

INTERVENTIONS:
Drug: aminolevulinic acid — Given orally
  Other Names: δ-Aminolevulinic acid Hydrochloride; 5-Amino-4-oxopentanoic acid Hydrochloride; 5-Aminolaevulinic acid Hydrochloride
Procedure: Surgical Resection — Surgical resection - 6 biopsies from 3 fluorescent regions

SUMMARY:
RATIONALE: Imaging procedures that use aminolevulinic acid (ALA) may help find and diagnose residual tumor in participants with grade IV malignant astrocytoma who are undergoing surgery to remove the tumor.

PURPOSE: Our primary long-term goal is to improve the completeness of surgical resection of malignant brain tumor through image- guided fluorescence localization. We hypothesize that the use of qualitative fluorescence imaging and point PpIX concentration quantification will enable more complete tumor resection than normal direct (i.e., white light) visualization, and thereby improve participant survival.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess 2 doses of 5-ALA, 10kg/mg and 20kg/mg, to determine the optimum ALA dose in terms of both sensitivity and specificity for residual tumor. We will compare residual tumor detection by both in vivo qualitative and quantitative fluorescence imaging using histology of the biopsied tissue as the gold standard.

Secondary

* Assess the correlation between the recorded in vivo qualitative assessment of fluorescence signal from the neurosurgeon with the post-surgical (i.e., ex vivo) absolute PpIX concentration detected both intraoperatively and in ex vivo tissue biopsies.

Tertiary

* To determine the association between the presence of fluorescence in the surgical cavity and the post-operative image enhancement on MRI. This includes the relationship between the amount and location of residual tumor detected by fluorescence, PpIX concentration, and intra-operative frameless stereotaxy following maximal resection versus the amount and location of tumor imaged post-operatively via CT and/or MRI.

OUTLINE: This study will enroll evaluable participants undergoing surgical resection of malignant, grade IV gliomas in both of two groups: those with , newly diagnosed GBM and those with recurrent GBM. Participants in each group (primary vs recurrent GBM) will be randomized to one of 2 levels of ALA dose (10 and20 mg/kg) to be given orally at 6 hours prior to anticipated midpoint of surgery.

Participants who have consented to this protocol will be randomly assigned to one of two ALA dose groups. Randomization will be stratified by whether the tumor is newly diagnosed (i.e. de novo) or recurrent. The data center will prepare sealed, opaque envelopes with the randomized assignment to ALA dose and administration time and notify the pharmacy of the trial site so that so that the correct ALA dose can be prepared.

* Arm I: Newly diagnosed GBM participants receive oral aminolevulinic acid(10mg/kg)at 6 hours before the midpoint of surgery.
* Arm II: Newly diagnosed GBM participants receive oral aminolevulinic acid (20mg/kg)at 6 hours before the midpoint of surgery.
* Arm III: Recurrent GBM participants receive oral aminolevulinic acid (10mg/kg)at 6 hours before the midpoint of surgery.
* Arm IV: Recurrent GBM participants receive oral aminolevulinic acid (20mg/kg)at 6 hours before the midpoint of surgery.

For both participants with new and recurrent disease, biopsies will be taken at up to six sites identified by the surgeon: in the tumor center, tumor edge, area surrounding the tumor (if safe), areas seen to fluoresce intraoperatively and an area with MR enhancement outside the tumor region (if this can be accomplished safely). Prior to collecting these biopsies readings will be taken at the biopsied location with the PpIX point probe by the surgeon. For each of the 6 biopsies, they will be divided into 3 parts and distributed for further analysis as follows: one portion will be sent to the pathologist for assessment of tumor percentage, one portion will be evaluated by the Division of Biophysics at the University of Toronto for PpIX concentration and the other for assessment of fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Tumor Pathology: Newly diagnosed or recurrent malignant gliomas WHO grade IV
* Location: Supratentorial
* Resection: Tumor must be judged suitable for resection on the basis of imaging studies.
* Consent: Participants must be able to give written, informed consent as approved by the local IRB
* Newly Diagnosed Tumors: Participants with newly diagnosed Grade IV glioma who have had not been previously treated with cranial radiation therapy
* Recurrent Tumors: Participants with recurrent Grade IV gliomas who have failed cranial radiation therapy

Exclusion Criteria:

* Pregnant women or those who are breast feeding
* Individuals with history of cutaneous photosensitivity, porphyria, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis
* Individuals with history of liver disease in last 12 months
* Individuals with AST, ALT, ALP, or bilirubin >2.5x normal upper limit any time during the previous 2 months
* Individuals with plasma creatinine>180 μmol/L
* Individuals who are unable to comply with photosensitivity precautions
* Individuals without a grade IV glioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
Assess 2 doses of 5-ALA | 6 hours before midpoint of surgery
  This clinical trial has ALA dose at 2 levels (10 and 20 mg/kg) and ALA administration time at 1 time point (6h). During surgery, the intraoperative fluorescence observations and PpIX concentration measurements will be taken by the surgeon. The second part of each biopsy will have the PpIX concentration determined.

SECONDARY OUTCOMES:
Correlation between intensity of in vivo fluorescence and the pathologist's quantification of tumor in biopsy specimens (e.g., percentage of tumor present) as measured by PpIX concentration and intra-operative fluorescence intensity | Quantitative fluorescence imaging of tumor tissue and normal tissue at approximately the midpoint of surgery and then after maximal resection of the tumor.
  readings will be taken at the biopsied location with the PpIX point probe by the surgeon.
Correlation between the amount and location of residual tumor detected intraoperatively by fluorescence imaging and frameless stereotaxy after maximal resection and the post-operative image enhancement on CT scan and/or MRI | Tumor tissue samples are obtained at the same two timepoints (the midpoint of surgery and then after maximal resection of the tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sloan, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT00752323/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT00752323/ICF_001.pdf